CLINICAL TRIAL: NCT00544648
Title: A Phase I/II Study of Nab-Paclitaxel and Carboplatin With Concurrent Radiation Therapy for Unresectable Stage III Non-Small-Cell Lung Cancer (NSCLC)
Brief Title: Ph I/II Nab-Paclitaxel & Carboplatin w/Concurrent Radiation Therapy for Unresectable Stg III NSCLC
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Ph I completed. Funding became unavailable causing Ph II to cease after two patients were enrolled.
Sponsor: Vanderbilt-Ingram Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Vicki Keedy, MD, Assistant Professor of Medicine; Clinical Director, Sarcoma Program; Medical Director, Clinical Trials Shared Resource; Medical Oncologist, Vanderbilt-Ingram Cancer Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: VICC THO 0746; P30CA068485 (NIH); VU-VICC-THO-0746
Record Dates: First submitted 2007-10-13; First posted 2007-10-16 (Estimated); Results first posted 2014-06-09 (Estimated); Last update posted 2014-06-09 (Estimated); Status verified 2014-05

CONDITIONS: Lung Cancer
Keywords: stage IV non-small cell lung cancer; stage IIIB non-small cell lung cancer
MeSH Terms: conditions — Lung Neoplasms; Carcinoma, Non-Small-Cell Lung | interventions — Carboplatin; 130-nm albumin-bound paclitaxel; Taxes; Albumin-Bound Paclitaxel; Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Treatment (Experimental): nab-paclitaxel+ carboplatin + radiation
  Interventions: Drug: carboplatin; Drug: nab-paclitaxel; Radiation: Radiation therapy

INTERVENTIONS:
Drug: carboplatin — (AUC 2) through a vein over 30 minutes following nab-paclitaxel, once per week x 7 weeks
  Other Names: Paraplatin
Drug: nab-paclitaxel — Phase I: beginning at 40 mg/m2 through a vein over 30 minutes once per week x 7 weeks Phase II: Maximum tolerated dose through a vein over 30 minutes once per week x 7 weeks
  Other Names: paclitaxel albumin-stabilized nanoparticle formulation; Abraxane
Radiation: Radiation therapy — 3D conformal radiotherapy or Intensity-Modulated Radiation Therapy (IMRT), 2.0 Gy per day x 5 days per week for 33 days during Weeks 1-7 ; Total Dose = 66 Gy

SUMMARY:
RATIONALE: Drugs used in chemotherapy, such as carboplatin, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Radiation therapy uses high-energy x-rays to kill tumor cells. Nab-paclitaxel (paclitaxel albumin-stabilized nanoparticle formulation) may make tumor cells more sensitive to radiation therapy. Giving nab-paclitaxel together with radiation therapy and carboplatin may kill more tumor cells.

PURPOSE: This phase I/II trial is studying the side effects and best dose of giving nab-paclitaxel together with carboplatin and radiation therapy and to see how well it works in treating patients with stage III non-small-cell lung cancer that cannot be removed by surgery.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* To determine the maximum tolerated dose of nab-paclitaxel when combined concurrently with carboplatin and radiation followed by two courses of nab-paclitaxel carboplatin as consolidation. (Phase I)
* To evaluate the progression-free survival in patients with stage III unresectable non-small cell lung cancer treated with nab-paclitaxel, carboplatin, and radiotherapy followed by two courses of nab-paclitaxel with carboplatin as consolidation. (Phase II)

Secondary

* To assess safety and tolerability and identify dose-limiting toxicities in patients receiving nab-paclitaxel combined concurrently with carboplatin and radiotherapy. (Phase I)
* To assess progression-free survival, response rates, and survival. (Phase I)
* To assess overall survival and response rates in all patients treated on this study. (Phase II)
* To assess the safety and tolerability of patients receiving nab-paclitaxel combined concurrently with carboplatin and radiotherapy followed by two courses of nab-paclitaxel/carboplatin as consolidation. (Phase II) OUTLINE: This is a multicenter study.
* Phase I:

  * Concurrent chemoradiotherapy: Patients receive escalating doses of nab-paclitaxel IV over 30 minutes and carboplatin IV over 30 minutes on days 1, 8, 15, 22, 29, 36, and 43. They also receive conformal radiotherapy once daily 5 days a week on days 1-5 in weeks 1-7. Patients are evaluated between weeks 8-10. Patients with disease progression are removed from study. Patients with stable disease, partial response, or complete response proceed to consolidation chemotherapy 3 weeks after completion of chemoradiotherapy.
  * Consolidation chemotherapy: Patients receive nab-paclitaxel IV over 30 minutes on days 1, 8, and 15 and carboplatin IV over 30 minutes on day 1. Treatment repeats ever 21 days for up to 2 courses.
* Phase II: Patients receive concurrent chemoradiotherapy at the Maximum Tolerated Dose (MTD) of nab-paclitaxel followed by consolidation chemotherapy as in phase I.

After completion of study treatment, patients are followed at 2 months, every 3 months for 2 years, every 4 months for 2 years, and then every 6 months thereafter.

PROJECTED ACCRUAL: A total of 98 patients (15 patients for phase I and 83 patients for phase II) will be accrued for this study.

ELIGIBILITY:
Inclusion Criteria for Phase I and Phase II Patients:

* Patients must voluntarily sign and date an informed consent before the initiation of any study procedures
* Patients must have non-metastatic, inoperable, Stage IIIA or IIIB histologically or cytologically documented NSCLC without evidence of malignant pleural effusion
* Patients must not have received any prior systemic chemotherapy, thoracic radiotherapy or surgical resection for treatment of NSCLC
* Patients must have at least one site of unidirectionally measurable disease as defined by Response Evaluation in Solid Tumors (RECIST) criteria
* Patients must be ≥ 3 weeks from a formal exploratory thoracotomy
* Patients must have a Radiation Oncology and Medical Oncology consult and approval prior to study entry
* Patients must be ≥ 18 years of age
* Patients must have an Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1
* Women of childbearing potential must have a negative baseline serum pregnancy or a negative urine pregnancy test within 7 days prior to Week 1, Day 1 and must not be breast feeding.
* Women of childbearing potential and men with a sexual partner of child bearing potential must use an effective method of contraception beginning prior to study entry, for the duration of the study participation and for a minimum of 3 months after the last dose of chemotherapy.
* Patients must have adequate hepatic, renal, lung and bone marrow function as defined below:

  * Absolute neutrophil count (ANC) ≥1,500/mm3
  * Hemoglobin ≥ 9.0 gm/dL
  * Serum Creatinine ≤1.5mg/dl
  * Platelets > 100,000/mm3
  * Total bilirubin ≤ upper limit of normal
  * AST and ALT < 2.5 X upper limit of normal
  * Alkaline phosphatase < 2.5 X upper limit of normal
  * Calculated CrCl > 45 ml/min (via Cockroft-Gault formula)
  * Forced expiratory volume in 1 second (FEV 1) > 800 ml

Exclusion Criteria for Phase I and Phase II Patients:

* Known hypersensitivity to carboplatin or nab-paclitaxel
* Peripheral neuropathy Grade ≥ 2
* Wet stage IIIB (documented malignant pleural effusion) or stage IV NSCLC
* Previous chemotherapy or radiation therapy to the chest
* Any concomitant malignancy or brain metastasis
* Any uncontrolled, clinically significant medical or psychiatric disorder
* Pregnant or nursing women
* A greater than or equal to 10% weight loss over the past 3 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2007-11; Primary Completion 2014-04 (Actual); Study Completion 2014-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Vicki Keedy, MD, Principal Investigator — Vanderbilt-Ingram Cancer Center
Locations (6):
- United States (6):
  - Purchase Cancer Group - Paducah, Paducah, Kentucky
  - Oregon Health Sciences University, Portland, Oregon
  - Erlanger Cancer Center at Erlanger Hospital - Baroness, Chattanooga, Tennessee
  - Vanderbilt-Ingram Cancer Center - Cool Springs, Nashville, Tennessee
  - Vanderbilt-Ingram Cancer Center at Franklin, Nashville, Tennessee
  - Vanderbilt-Ingram Cancer Center, Nashville, Tennessee

REFERENCES:
- [Derived] Lammers PE, Lu B, Horn L, Shyr Y, Keedy V. nab-Paclitaxel in Combination With Weekly Carboplatin With Concurrent Radiotherapy in Stage III Non-Small Cell Lung Cancer. Oncologist. 2015 May;20(5):491-2. doi: 10.1634/theoncologist.2015-0030. Epub 2015 Apr 6. PMID 25845992

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients were recruited from November 2007 through September 2011
Pre-assignment Details: Twenty-two patients signed consent on this study, nine of which were ineligible to receive treatment.
Groups:
- Phase I: Nab-paclitaxel in mg/m2 of nab-paclitaxel in combination with carboplatin AUC 2 weekly for 7 weeks with concurrent radiotherapy
- Phase II: MTD of Nab-paclitaxel in mg/m2 in combination with carboplatin AUC 2 with concurrent radiotherapy weekly for 7 weeks. Responding patients will be treated with consolidation chemotherapy of nab-paclitaxel 100 mg/m2 weekly for 3 weeks every 21 days followed by carboplatin on day 1 of each cycle. One cycle is 21 days. Patients receive 2 cycles of this consolidation chemotherapy.
Period: Overall Study
Arm/Group | Phase I | Phase II
Started | 11 | 2
Completed | 8 | 1
Not Completed | 3 | 1
Not completed — Withdrawal by Subject | 1 | 0
Not completed — Adverse Event | 1 | 1
Not completed — progression of disease | 1 | 0

BASELINE CHARACTERISTICS:
Population: Consented patients
Groups:
- Total: Total of all reporting groups
Arm/Group | Phase I | Phase II | Total
Number analyzed (Participants) | 11 | 2 | 13
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 4 | 2 | 6
  >=65 years | 7 | 0 | 7
Age, Continuous [Mean (Standard Deviation); unit: years] | 63 (9) | 56 (4) | 59 (16)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 1 | 3
  Male | 9 | 1 | 10
Region of Enrollment [Number; unit: participants]
  United States | 11 | 2 | 13

OUTCOME MEASURES:

1. Primary Outcome: Maximum Tolerated Dose of Nab-paclitaxel When Combined Concurrently With Carboplatin and Radiation (Phase I)
Description: The highest dose in milligrams per meter of body surface squared (mg/m2) of nab-paclitaxel in combination with carboplatin while maintaining tolerability. Cohorts of 3-6 patients received escalating doses of nab-paclitaxel in combination with carboplatin until the maximum tolerated dose (MTD) was achieved. The MTD is defined as the dose preceding that at which 2 or more of 6 patients experience dose-limiting toxicity (DLT) during the initial cycle of therapy. DLTs per Common Toxicity Criteria v 3.0: recurring non-hematological (except esophagitis) > Grade 2, non-hematological or esophagitis > Grade 3 toxicities that are symptomatically unacceptable to patient and result in treatment delay for > 2 weeks, persistent toxicity resulting in treatment delay for > 2 weeks.
Time Frame: 7 weeks
Population: MTD based on clinical performance of those patients who received the study drug. One patient withdrew before receiving treatment. No formal statistical analysis, such as hypothesis testing, was performed.
Measure: Number; unit: mg/m2
Arm/Group | Phase I
Number analyzed (Participants) | 10
mg/m2 | 40

2. Primary Outcome: Progression-free Survival (Phase II)
Description: Estimated probable duration of life without disease progression, from on-study date to earlier of progression date, or date of death from any cause, using the Kaplan-Meier method with censoring (see Analysis Population Description for additional details). Disease progression is defined by Response Evaluation in Solid Tumors (RECIST) v.1.1: >= 20% increase in sum of the longest diameter of target lesions, unequivocal progression of non-target lesions, or appearance of new lesions
Time Frame: On-study to lesser of date of progression or date of death from any cause (assessed up to 2 years)
Population: All patients are included in the analysis on intention-to-treat basis. Analysis is by Kaplan-Meier method, where either death or progression is an event, with censoring for non-progressed, non-expired patients at greater of off-study date or last known date alive.
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Phase II
Number analyzed (Participants) | 2
days | 126 [126 to NA] — Upper bound of the 95% confidence interval could not be estimated because of lack of events and patients

3. Secondary Outcome: Progression-free Survival (Phase I)
Description: as for outcome 2
Time Frame: On-study to lesser of date of progression or date of death from any cause (assessed up to 2 years)
Population: as for outcome 2
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Phase I
Number analyzed (Participants) | 11
days | 231 [120 to 492]

4. Secondary Outcome: Overall Survival (Phase I)
Description: Estimated probable duration of life from on-study date to date of death from any cause, using Kaplan-Meier method with censoring (see Analysis Population Description for additional details).
Time Frame: On-study date to date of death from any cause (assessed up to 2 years)
Population: All patients are included in the analysis on intention-to-treat basis. Analysis is by Kaplan-Meier method, where death is an event, with censoring for non-expired patients at greater of off-study date or last known alive date.
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Phase I
Number analyzed (Participants) | 11
days | 575 [257 to NA] — Upper bound of the 95% confidence interval could not be estimated due to lack of events

5. Secondary Outcome: Response (Phase I)
Description: Number of patients in each response category, per Response Evaluation in Solid Tumors (RECIST) v.1.1: complete response (CR), disappearance of target lesions; partial response (PR) >=30% decrease in sum of longest diameter (LD) of target lesions; progressive disease (PD), >=20% increase in sum of LD of target lesions or appearance of new lesions; stable disease (SD), insufficient change in target lesions or new lesions to qualify as either PD or PR. Patients are categorized according to the best response achieved prior to occurrence of progressive disease, where best response hierarchy is CR>PR>SD>PD.
Time Frame: On-treatment date to date of progressive disease (assessed up to 2 years)
Population: All patients with best overall response data; patients are excluded if best overall response data is missing (0) or if the patient is non-evaluable for best overall response (n = 1)
Measure: Number; unit: participants
Arm/Group | Phase I
Number analyzed (Participants) | 10
participants
  Complete response | 0
  Partial response | 9
  Stable disease | 1
  Progressive disease | 0

6. Secondary Outcome: Number of Patients With Each Worst Grade Toxicity (Phase I)
Description: Count of patients according to the worst-grade toxicity (WGT) experienced by each, where worst-grade toxicity is per NCI common toxicity criteria: Grade 1, mild; Grade 2, moderate; Grade 3, severe; Grade 4, life-threatening; Grade 5, death.
Time Frame: On-study date to 30 days following final dose of study drug
Population: Total number of patients reported with any toxicity. One patient did not experience toxicity.
Measure: Number; unit: participants
Groups:
- Phase I: Nab-paclitaxel in mg/m2 of nab-paclitaxel in combination with carboplatin AUC 2 with concurrent radiotherapy
Arm/Group | Phase I
Number analyzed (Participants) | 10
participants
  Number of patients with worst Grade 1 toxicity | 0
  Number of patients with worst grade 2 toxicity | 2
  Number of patients with worst grade 3 toxicities | 5
  Number of patients with worst grade 4 toxicity | 3
  Number of patients with worst grade 5 toxicity | 0

7. Secondary Outcome: Overall Survival (Phase II)
Description: Estimated probable duration of life from on-study date to date of death from any cause, using Kaplan-Meier method with censoring (see Analysis Population Description for additional details. Too few patients were enrolled in the Phase II arm for an analysis of overall survival
Time Frame: Time Frame: date on study to date of death from any cause or last known date alive
Population: Too few patients were enrolled in the Phase II arm for an analysis of overall survival
Arm/Group | Phase II
Number analyzed (Participants) | 0

8. Secondary Outcome: Number of Patients With Each Worst Grade Toxicity (Phase II)
Description: The number of patients with worst-grade toxicity at each of five grades following NCI Common Toxicity Criteria: 1 = mild, 2 = moderate, 3 = severe, 4 = life-threatening, disabling, 5 = death
Time Frame: at 16 weeks
Population: Treated patients who experienced a toxicity.
Measure: Number; unit: participants
Arm/Group | Phase II
Number analyzed (Participants) | 2
participants
  Number of patients with worst grade 1 toxicity | 0
  Number of patients with worst grade 2 toxicity | 1
  Number of patients with worst grade 3 toxicity | 1
  Number of patients with worst grade 4 toxicity | 0
  Number of patients with worst grade 5 toxicity | 0

9. Secondary Outcome: Response (Phase II)
Description: as for outcome 5
Time Frame: On-treatment date to date of progressive disease (assessed up to 2 years)
Population: All patients with best overall response data; patients are excluded if best overall response data is missing (n = 0) or if the patient is non-evaluable for best overall response (n = 1)
Measure: Number; unit: participants
Arm/Group | Phase II
Number analyzed (Participants) | 1
participants
  Complete response | 0
  Partial response | 1
  Stable disease | 0
  Progressive disease | 0

10. Other Pre Specified Outcome: Secreted Protein Acidic and Rich in Cysteine (SPARC) Gene Expression
Description: Secreted protein acidic and rich in cysteine (SPARC) gene expression in tumor specimens.
Time Frame: On receipt of tumor tissue blocks
Population: Investigators elected not to perform this analysis.
Groups:
- Phase I and Phase II: Phase I-Nab-paclitaxel in mg/m2 in combination with carboplatin AUC 2 with concurrent radiotherapy weekly for 7 weeks. Responding patients will be treated with consolidation chemotherapy of nab-paclitaxel 100 mg/m2 weekly for 3 weeks every 21 days followed by carboplatin on day 1 of each cycle. One cycle is 21 days. Patients receive 2 cycles of this consolidation chemotherapy.
  Phase II-MTD Nab-paclitaxel in mg/m2 in combination with carboplatin AUC 2 with concurrent radiotherapy weekly for 7 weeks. Responding patients will be treated with consolidation chemotherapy of nab-paclitaxel 100 mg/m2 weekly for 3 weeks every 21 days followed by carboplatin on day 1 of each cycle. One cycle is 21 days. Patients receive 2 cycles of this consolidation chemotherapy.
  Phase II-
Arm/Group | Phase I and Phase II
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: This study began November 2007 through September 2011. Data were collected through April 2013.
Description: One patient withdrew before receiving treatment
Groups:
- Phase I: Nab-paclitaxel in mg/m2 in combination with carboplatin AUC 2 with concurrent radiotherapy weekly for 7 weeks. Responding patients will be treated with consolidation chemotherapy of nab-paclitaxel 100 mg/m2 weekly for 3 weeks every 21 days followed by carboplatin on day 1 of each cycle. One cycle is 21 days. Patients receive 2 cycles of this consolidation chemotherapy.
Arm/Group | Phase I | Phase II
Serious Adverse Events (participants affected / at risk) | 5/10 | 1/2
Other Adverse Events (participants affected / at risk) | 10/10 | 2/2
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Phase I (N=10) | Phase II (N=2)
hemoglobin (Blood and lymphatic system disorders) | 1 (2) | 0 (0)
neutrophils (Blood and lymphatic system disorders) | 4 (4) | 0 (0)
platelets (Blood and lymphatic system disorders) | 3 (3) | 0 (0)
radiation dermatitis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
hyponatremia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
thrombosis (Vascular disorders) | 2 (2) | 0 (0)
febrile neutropenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
digoxin toxicity (Cardiac disorders) | 1 (1) | 0 (0)
sore throat (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
fever in the absence of neutropenia (defined as ANC < 1.0 x 10e9/L) (General disorders) | 1 (1) | 0 (0)
hypotension (Cardiac disorders) | 1 (1) | 0 (0)
hypoxia (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
International Ratio of prothrombin time (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
speech impairment (Nervous system disorders) | 1 (1) | 0 (0)
atrial fibrillation (Cardiac disorders) | 1 (1) | 0 (0)
sinus tachycardia, probably related to pneumonia (Cardiac disorders) | 0 (0) | 1 (1)
pain-chest, thorax NOS (General disorders) | 0 (0) | 1 (1)
dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
tachypnea, probably related to pneumonia (Cardiac disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Phase I (N=10) | Phase II (N=2)
hemoglobin (Blood and lymphatic system disorders) | 10 (24) | 2 (6)
leukocytes (total WBC) (Blood and lymphatic system disorders) | 4 (13) | 1 (6)
neutrophils/granulocytes (ANC/ANG) (Blood and lymphatic system disorders) | 2 (6) | 1 (1)
platelets (Blood and lymphatic system disorders) | 4 (12) | 1 (4)
blood/bone marrow-other (Blood and lymphatic system disorders) | 3 (5) | 0 (0)
nausea (Gastrointestinal disorders) | 4 (4) | 2 (6)
dehydration (Gastrointestinal disorders) | 3 (3) | 1 (2)
diarrhea (Gastrointestinal disorders) | 3 (4) | 1 (2)
anorexia (Gastrointestinal disorders) | 3 (3) | 0 (0)
vomiting (Gastrointestinal disorders) | 1 (1) | 2 (5)
constipation (Gastrointestinal disorders) | 2 (2) | 0 (0)
esophagitis (Gastrointestinal disorders) | 2 (2) | 0 (0)
mucositis/stomatitis (functional/symptomatic)-esophagus (Gastrointestinal disorders) | 1 (1) | 1 (2)
dysphagia (Gastrointestinal disorders) | 1 (2) | 0 (0)
flatulence (Gastrointestinal disorders) | 1 (1) | 0 (0)
heartburn/dyspepsia (Gastrointestinal disorders) | 1 (1) | 0 (0)
mucositits/stomatitis (functional/symptomatic) oral cavity (Gastrointestinal disorders) | 1 (1) | 0 (0)
taste alteration (Gastrointestinal disorders) | 1 (1) | 0 (0)
fatigue (General disorders) | 9 (10) | 2 (2)
constitutional symptoms-other (General disorders) | 4 (8) | 1 (4)
insomnia (Psychiatric disorders) | 3 (4) | 0 (0)
fever in the absence of neutropenia, where neutropenia is defined as ANC < 1.0 x 10e9/L (General disorders) | 3 (3) | 0 (0)
sweating (General disorders) | 2 (2) | 0 (0)
hypomagnesemia (Metabolism and nutrition disorders) | 7 (9) | 1 (2)
hyperglycemia (Metabolism and nutrition disorders) | 10 (13) | 1 (3)
ALT, SGPT (serum glutamic pyruvic transaminase) (Metabolism and nutrition disorders) | 2 (3) | 1 (3)
metabolic/laboratory-other (Metabolism and nutrition disorders) | 2 (2) | 1 (1)
hypophosphatemia (Metabolism and nutrition disorders) | 2 (2) | 1 (1)
hypokalemia (Metabolism and nutrition disorders) | 3 (4) | 0 (0)
hyponatremia (Metabolism and nutrition disorders) | 1 (2) | 1 (4)
hypoalbuminemia (Metabolism and nutrition disorders) | 2 (3) | 0 (0)
AST, SGOT (serum glutamic oxaloacetic transaminase (Metabolism and nutrition disorders) | 1 (1) | 1 (2)
alkaline phosphatase (Metabolism and nutrition disorders) | 1 (2) | 0 (0)
hyperbilirubinemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
hypocalcemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
creatinine (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
hypermagnesemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
pain-chest wall (Musculoskeletal and connective tissue disorders) | 3 (3) | 0 (0)
pain-back (Musculoskeletal and connective tissue disorders) | 2 (2) | 1 (1)
pain-head/headache (Nervous system disorders) | 2 (2) | 0 (0)
pain-throat, larynx (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
pain-chest, thorax (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
pain-extremity, limb (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
pain-joint (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
burn (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0)
dermatology, skin-other (Skin and subcutaneous tissue disorders) | 1 (2) | 1 (2)
dry skin (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0)
rash-dermatitis, radiation (Skin and subcutaneous tissue disorders) | 1 (4) | 0 (0)
alopecia (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
pruritis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
rash/desquamation (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
rash-acne/acneiform (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
cough (Respiratory, thoracic and mediastinal disorders) | 6 (6) | 1 (2)
dyspnea (Respiratory, thoracic and mediastinal disorders) | 5 (5) | 0 (0)
hypoxia (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
pneumonia/pulmonary infiltrates (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
febrile neutropenia (ANC < 1.0 x 10e9/L, fever >= 38.5 degrees Celsius (Infections and infestations) | 1 (1) | 0 (0)
infection-upper airway with Grade 3 or 4 neutrophils, ANC < 1.0 x 10e9/L (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
infection-other (Infections and infestations) | 1 (1) | 0 (0)
infection-bladder, normal ANC or Grade 1 or 2 neutrophils (Renal and urinary disorders) | 1 (1) | 0 (0)
infection-sinus, normal ANC or Grade 1 or 2 neutrophils (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
infection-stomach, with normal ANC or Grade 1 or 2 neutrophils (Gastrointestinal disorders) | 1 (1) | 0 (0)
dizziness (Nervous system disorders) | 2 (2) | 0 (0)
anxiety (Psychiatric disorders) | 1 (1) | 0 (0)
neurology-other (Nervous system disorders) | 1 (1) | 0 (0)
tremor (Nervous system disorders) | 1 (1) | 0 (0)
hypotension (Cardiac disorders) | 2 (2) | 0 (0)
cardiac general-other (Cardiac disorders) | 1 (1) | 0 (0)
hot flashes/flushes (Endocrine disorders) | 1 (1) | 0 (0)
hemorrhage-nose (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
edema-limb (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
erectile dysfunction (Reproductive system and breast disorders) | 1 (1) | 0 (0)
gastrointestinal other (Gastrointestinal disorders) | 0 (0) | 1 (1)
hypercalcemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
pain-bone (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
pain-cardiac (Cardiac disorders) | 0 (0) | 1 (1)
Infection with normal ANC or grade 1 or 2 neutrophils (Infections and infestations) | 0 (0) | 1 (1)
Infection with unknown ANC-pneumonia (Infections and infestations) | 0 (0) | 1 (1)

LIMITATIONS AND CAVEATS:
This Phase I/II study progressed into Phase II, but terminated shortly thereafter due to lack of funding.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes